CLINICAL TRIAL: NCT05599893
Title: Role of Tele-physical Therapy Training on Glycemic Control, Pulmonary Function, Physical Fitness, and Health-related Quality of Life in Patients With Type 2 Diabetes Mellitus Following COVID-19 Infection - a Randomized Controlled Trial.
Brief Title: Role of Tele-physical Therapy in Patients With Type 2 Diabetes Mellitus Following COVID-19 Infection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/021/085
Record Dates: First submitted 2022-10-28; First posted 2022-10-31 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus; COVID-19
MeSH Terms: conditions — Diabetes Mellitus, Type 2; COVID-19

STUDY DESIGN:
Intervention Model Description: The participants were randomized into either of these two groups in 1:1 ratio through two block (block size 12-15) simple random sampling method. Tele - physical therapy group (TPG; n = 68) and a control intervention group (CIG; n = 68). To ensure allocation concealment, an independent therapist randomly picked up an envelope that contained patient information, in a blinded fashion and segregated the patient into either of these two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The treating therapists could not be blinded due to practical feasibility. Assessing therapists measured the outcomes of each participant at each interval without knowing the group allocation. Participants were also blinded by requesting them not to disclose their allocation to the assessing therapists and co-participants at any time during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele - physical therapy group (Experimental): Participants in the tele-physical therapy group underwent tele-physical therapy sessions which includes an internet-based video conference under the supervision of physical therapists. Before commencing training, warm-up exercises involving upper and lower extremity joint movements were performed for 10 times. During the first and second weeks, the third and fourth weeks, the fifth and sixth weeks and the seventh and eighth weeks, the exercises were performed 10-15, 15-20, 20-25 and 25-30 times per session, respectively. Each session lasted for 10 minutes of warm-up, 60 minutes of training and 10 minutes of a cool-down phase. The participants in the tele physical therapy group received training four times a week, for 8 weeks, each session lasted for 60 minutes.
  Interventions: Other: Tele physical therapy
- Control intervention group (Active Comparator): During the first visit, participants in the control intervention group (CIG) received patient education for 10 minutes from physical therapists and also received a pamphlet containing these instructions in written form. They were informed to do their normal daily activities, avoid sedentary lifestyle, perform regular physical activities such as household activities, maintain balance diet and have 6-8 hours of sleep per day.
  Interventions: Other: Patient educationa and Conventional exercises

INTERVENTIONS:
Other: Tele physical therapy — Before commencing training, warm-up exercises involving upper and lower extremity joint movements were performed for 10 times. During the first and second weeks, the third and fourth weeks, the fifth and sixth weeks and the seventh and eighth weeks, the exercises were performed 10-15, 15-20, 20-25 and 25-30 times per session, respectively. Each session lasted for 10 minutes of warm up, 60 minutes of training and 10 minutes of cool down phase. The participants in the TPG received training four times a week, for 8 weeks, each session lasted for 60 minutes.
  Arms: Tele - physical therapy group
Other: Patient educationa and Conventional exercises — They were informed to do their normal daily activities, avoid a sedentary lifestyle, perform regular physical activities such as household activities, maintain a balanced diet and have 6-8 hours of sleep per day.
  Arms: Control intervention group

SUMMARY:
Diabetes mellitus (DM) is a chronic metabolic disease where the body is unable to metabolize carbohydrates properly either due to a lack of insulin production or abnormal insulin function. In recent times, it has been considered a global healthcare concern because of its high prevalence rate (9.2 %) and other associated health consequences. After being infected with Coronavirus disease-2019 (COVID-19), the Type 2 Diabetes mellitus (T2DM) sufferer experiences the following symptoms; reduced exercise tolerance, decreased muscle strength, altered respiratory functions, cognitive impairments and abnormal psychosomatic behaviour, which affects the overall well-being of the patient. To prevent or delay these clinical features and the associated consequences of type 2 Diabetes mellitus, the regular body works out and physical training is suggested either alone or in combination with diet modification. In this study, we tested the hypothesis that 12 months of supervised tele-physical therapy can positively influence patients with type 2 diabetes mellitus following COVID-19 infection. The reports of the study would be helpful for the clinicians and the physical therapists to make this as evidence for using tele-physical therapy in type 2 Diabates mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18-60 years of age and being diagnosed with COVID-19 with mild dyspnea and type 2 DM and the ability to use smart mobile phones were selected to be included in the study.

Exclusion Criteria:

* Participants who had neurological (radiculopathy, myelopathy and disc problems) and orthopedic problems, cardio-pulmonary diseases (stroke, hypertension and syncope), other metabolic and endocrinal problems, metastasis, pregnancy, taking analgesics or corticosteroids, any contra indications to physical exercises (fracture, instability, osteoporosis, arthropathy and neural symptoms) and cognitive and mental disorder were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic level | Baseline
  The hemoglobin A1C test, also known as HbA1c test. It is a simple blood test which measures the blood sugar levels of the participants.
Glycemic level | 8 weeks
  The hemoglobin A1C test, also known as HbA1c test. It is a simple blood test which measures the blood sugar levels of the participants.
Glycemic level | 6 months
  The hemoglobin A1C test, also known as HbA1c test. It is a simple blood test which measures the blood sugar levels of the participants.
Glycemic level | 12 months
  The hemoglobin A1C test, also known as HbA1c test. It is a simple blood test which measures the blood sugar levels of the participants.

SECONDARY OUTCOMES:
Forced Expiratory volume 1 | Baseline
  It measures the forced expiratory volume in the first second (FEV1) in litres
Forced Expiratory volume 1 | 8 weeks
  It measures the forced expiratory volume in the first second (FEV1) in litres
Forced Expiratory volume 1 | 6 months
  It measures the forced expiratory volume in the first second (FEV1) in litres
Forced Expiratory volume 1 | 12 months
  It measures the forced expiratory volume in the first second (FEV1) in litres
Forced vital capacity | Baseline
  It measures the forced vital capacity (FVC) in litres.
Forced vital capacity | 8 weeks
  It measures the forced vital capacity (FVC) in litres.
Forced vital capacity | 6 months
  It measures the forced vital capacity (FVC) in litres.
Forced vital capacity | 12 months
  It measures the forced vital capacity (FVC) in litres.
Forced vital capacity/Forced Expiratory volume 1 | Baseline
  It measures the forced expiratory volume1/forced vital capacity in percentage.
Forced vital capacity/Forced Expiratory volume 1 | 8 weeks
  It measures the forced expiratory volume1/forced vital capacity in percentage.
Forced vital capacity/Forced Expiratory volume 1 | 6 months
  It measures the forced expiratory volume1/forced vital capacity in percentage.
Forced vital capacity/Forced Expiratory volume 1 | 12 months
  It measures the forced expiratory volume1/forced vital capacity in percentage.
Maximum voluntary ventilation | Baseline
  It measures the maximum voluntary ventilation (MVV) in liters/minute.
Maximum voluntary ventilation | 8 weeks
  It measures the maximum voluntary ventilation (MVV) in liters/minute.
Maximum voluntary ventilation | 6 months
  It measures the maximum voluntary ventilation (MVV) in liters/minute.
Maximum voluntary ventilation | 12 months
  It measures the maximum voluntary ventilation (MVV) in liters/minute.
Peak exploratory flow | Baseline
  It measures the peak exploratory flow (PEF) in liters/second.
Peak exploratory flow | 8 weeks
  It measures the peak exploratory flow (PEF) in liters/second.
Peak exploratory flow | 6 months
  It measures the peak exploratory flow (PEF) in liters/second.
Peak exploratory flow | 12 months
  It measures the peak exploratory flow (PEF) in liters/second.
Physical fitness | Baseline
  It was measured with six-minute walk test ,which assess the functional exercise capacity of the participants. Higher the scores represent better results and the lower scores represent worst results.
Physical fitness | 8 weeks
  It was measured with six-minute walk test ,which assess the functional exercise capacity of the participants. Higher the scores represent better results and the lower scores represent worst results.
Physical fitness | 6 months
  It was measured with six-minute walk test ,which assess the functional exercise capacity of the participants. Higher the scores represent better results and the lower scores represent worst results.
Physical fitness | 12 months
  It was measured with six-minute walk test ,which assess the functional exercise capacity of the participants. Higher the scores represent better results and the lower scores represent worst results.
Health related quality of life | Baseline
  It was evaluated with the Short Form Health Survey-12 (SF-12). Higher the scores represent better results and the lower scores represent worst results.
Health related quality of life | 8 weeks
  It was evaluated with the Short Form Health Survey-12 (SF-12). Higher the scores represent better results and the lower scores represent worst results.
Health related quality of life | 6 months
  It was evaluated with the Short Form Health Survey-12 (SF-12). Higher the scores represent better results and the lower scores represent worst results.
Health related quality of life | 12 months
  It was evaluated with the Short Form Health Survey-12 (SF-12). Higher the scores represent better results and the lower scores represent worst results.

CONTACTS AND LOCATIONS:
Locations (1):
- Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: After publication